CLINICAL TRIAL: NCT07324538
Title: A Randomized Controlled Trial Comparing the Immediate Effects of Manual and Verbal Cueing During Movement Control Training in Individuals With Chronic Non-Specific Low Back Pain
Brief Title: Immediate Effects of Manual and Verbal Cueing During Movement Control Training in Chronic Non-Specific Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Wendy Tzyy-Jiuan Wang, Professor, Department of Physical Therapy, National Yang Ming Chiao Tung University, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NYCU114229AE-S2
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Chronic Low Back Pain (Non-specific, Uncomplicated)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Cueing Followed by Verbal Cueing (Experimental)
  Interventions: Behavioral: Movement Control Training With Manual Cueing; Behavioral: Movement Control Training With Verbal Cueing
- Verbal Cueing Followed by Manual Cueing (Experimental)
  Interventions: Behavioral: Movement Control Training With Manual Cueing; Behavioral: Movement Control Training With Verbal Cueing

INTERVENTIONS:
Behavioral: Movement Control Training With Manual Cueing — Movement Control Training with Manual Cueing involves hands-on guidance provided by the therapist to enhance movement quality during standardized movement control training. Verbal instructions are used only to explain the movement sequence, while manuel guidance is primarily applied to facilitate movement quality.
  Manual cueing is delivered according to the individual's needs and may include the following strategies:
  1. Gentle and evenly distributed manual pressure is applied to provide postural support and enhance awareness of appropriate points of support during movement.
  2. Manuel guidance is used to assist joint alignment when suboptimal alignment is observed during task performance, with attention to maintaining balanced muscle tone.
  3. Joint approximation techniques are applied as needed to provide compressive and stabilizing input to the joints, commonly used in neuromuscular facilitation approaches, to enhance joint stability and sensory feedback during movement.
Behavioral: Movement Control Training With Verbal Cueing — Movement control training with verbal cueing involves the use of spoken instructions and verbal feedback provided by the therapist to facilitate movement quality during standardized movement control training. Physical contact is not used during the intervention.
  Verbal instructions are focused on key aspects of movement performance, including alignment and weight distribution, to support correct execution of the movement tasks. Examples of verbal cues include instructions such as maintaining the knee in a neutral position or directing attention to the distribution of load through the shoulder girdle during task performance.

SUMMARY:
Chronic non-specific low back pain is commonly associated with impaired movement control. Movement control training is often used in rehabilitation, and different cueing methods may influence how patients perform and learn movements.

The purpose of this randomized controlled trial is to compare the immediate effects of manual cueing and verbal cueing during movement control training in individuals with chronic non-specific low back pain. Participants will be randomly assigned to receive either manual cueing or verbal cueing during a standardized movement training session.

The study will examine immediate changes in movement control performance, perceived difficulty, and related clinical outcomes following the intervention. The results of this study may help clinicians better understand how different cueing strategies influence movement performance in people with chronic non-specific low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Clinically diagnosed chronic non-specific low back pain with symptoms lasting longer than 12 weeks
* Able to understand and comply with the assessment and intervention procedures

Exclusion Criteria:

* History of surgery involving the lower back or lower extremities
* Presence of neurological symptoms, such as paresthesia or numbness
* Signs or symptoms of nerve root compression
* History of surgery within the past 3 months
* History of cancer
* Presence of major medical or psychiatric disorders
* Presence of systemic inflammatory conditions
* Pregnancy
* Structural scoliosis
* Inability to walk or stand independently, or any condition deemed unsuitable for participation by the investigator
* Participation in any movement control exercise training within the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2026-11-15 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Movement Control Performance | Immediately before and immediately after each intervention period
  Movement control performance assessed using the Nine-Item Movement Control Test Battery, which evaluates movement quality during standardized functional movement tasks. Each item is scored according to predefined error-based criteria, and item scores are summed to produce a total score ranging from 0 to 93, with higher scores indicating poorer movement control performance.
Pain Intensity | Immediately before and immediately after each intervention period
  Pain intensity assessed using the Visual Analogue Scale (VAS), ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain imaginable, with higher scores indicating greater pain intensity.

SECONDARY OUTCOMES:
Perceived Difficulty Index | Immediately after each intervention period
  Perceived difficulty during movement performance assessed using the Perceived Difficulty Index (PDI). Participants rate the level of difficulty experienced during the movement tasks on a numeric rating scale ranging from 0 to 10, where 0 indicates no perceived difficulty and 10 indicates extreme difficulty, with higher scores indicating greater perceived difficulty.
Perceived Learning Effect | Immediately after each intervention period
  Perceived learning following each intervention session, assessed by the therapist using a numeric rating scale from 0 (no learning) to 10 (complete mastery of key movement principles).